CLINICAL TRIAL: NCT00679757
Title: The Prevalence and Implications of Obstructive Sleep Apnea in the Population of a Wound Center
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Dr. Rami Khayat, The Ohio State University
Other Study IDs: 2007H0242
Record Dates: First submitted 2008-05-15; First posted 2008-05-19 (Estimated); Last update posted 2010-06-10 (Estimated); Status verified 2010-06

CONDITIONS: Obstructive Sleep Apnea; Non-healing Wounds
Keywords: Sleep apnea; Obstructive sleep apnea; Wound healing; Non-healing wounds
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
This study is looking at the prevalence of sleep apnea in a wound center population. It uses both screening surveys and take home devices. Some measures of wound healing ability are being looked at as well.

DETAILED DESCRIPTION:
Patients with chronic non-healing wounds often have major co-morbidities such as diabetes and cardiovascular diseases [1]. Obstructive Sleep Apnea (OSA) is present in up to 24% of middle-aged adults [2], and is far more prevalent in patients with existing cardiovascular disease [3]. Patients with OSA are at increased risk of developing diabetes l [4]. OSA is an established cause of hypertension[5], and has an estimated prevalence of 40% in all patients with hypertension [6-8]. Similarly a strong association exists between OSA, coronary artery disease [6, 7] and stroke [8]. OSA may be present in over 50% of patients with heart failure [9]. Patients with chronic non-healing wounds stand to benefit from identification and treatment of severe co-morbidities such as OSA. Such identification and treatment of OSA will impact the survival of these patients [10, 11], and may also contribute to improved morbidity via impacting wound healing.

Several unexplored links exist between OSA and wound healing. OSA is a disorder of intermittent hypoxia and is associated with increased oxidative stress [12]. Humans with OSA and animal models of intermittent hypoxia developed impaired vascular function and nitric oxide deficiency. Patients with OSA have impaired endothelial function even in the absence of clinically apparent cardiovascular disease [13-15]. Increased sympathetic activity and episodic pressor response are well documented in OSA. Patients with OSA have increased vascular tone and baseline vasoconstriction [16]. Impaired vascular reactivity to hypoxia was also demonstrated in animal models exposed to 2 weeks of intermittent hypoxia[17]. Therefore, in patients with chronic non-healing wounds, OSA is likely to further complicate the healing process.

OSA as a disorder of oxidative stress and vascular impairment is most likely an important co-morbidity in patients with non-healing wounds. Other potential mechanisms of interaction are the inflammatory response associated with OSA

ELIGIBILITY:
Inclusion Criteria:

* OSU Wound Clinic Patient

Exclusion Criteria:

* Unable to complete survey
* Under 18yrs old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients of the OSU Wound Center
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2008-01; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Risk of having sleep apnea. | Immediate

SECONDARY OUTCOMES:
Wound healing ability. | Immediate

CONTACTS AND LOCATIONS:
Overall Officials: Rami N Khayat, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- [Background] Peivandi AA, Kasper-Konig W, Quinkenstein E, Loos AH, Dahm M. Risk factors influencing the outcome after surgical treatment of complicated deep sternal wound complications. Cardiovasc Surg. 2003 Jun;11(3):207-12. doi: 10.1016/s0967-2109(03)00006-1. PMID 12704330
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Javaheri S, Parker TJ, Liming JD, Corbett WS, Nishiyama H, Wexler L, Roselle GA. Sleep apnea in 81 ambulatory male patients with stable heart failure. Types and their prevalences, consequences, and presentations. Circulation. 1998 Jun 2;97(21):2154-9. doi: 10.1161/01.cir.97.21.2154. PMID 9626176
- [Background] Reichmuth KJ, Austin D, Skatrud JB, Young T. Association of sleep apnea and type II diabetes: a population-based study. Am J Respir Crit Care Med. 2005 Dec 15;172(12):1590-5. doi: 10.1164/rccm.200504-637OC. Epub 2005 Sep 28. PMID 16192452
- [Background] Young T, Peppard P, Palta M, Hla KM, Finn L, Morgan B, Skatrud J. Population-based study of sleep-disordered breathing as a risk factor for hypertension. Arch Intern Med. 1997 Aug 11-25;157(15):1746-52. PMID 9250236
- [Background] Peker Y, Carlson J, Hedner J. Increased incidence of coronary artery disease in sleep apnoea: a long-term follow-up. Eur Respir J. 2006 Sep;28(3):596-602. doi: 10.1183/09031936.06.00107805. Epub 2006 Apr 26. PMID 16641120
- [Background] Peker Y, Kraiczi H, Hedner J, Loth S, Johansson A, Bende M. An independent association between obstructive sleep apnoea and coronary artery disease. Eur Respir J. 1999 Jul;14(1):179-84. doi: 10.1034/j.1399-3003.1999.14a30.x. PMID 10489848
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Sin DD, Fitzgerald F, Parker JD, Newton G, Floras JS, Bradley TD. Risk factors for central and obstructive sleep apnea in 450 men and women with congestive heart failure. Am J Respir Crit Care Med. 1999 Oct;160(4):1101-6. doi: 10.1164/ajrccm.160.4.9903020. PMID 10508793
- [Background] Marin JM, Carrizo SJ, Vicente E, Agusti AG. Long-term cardiovascular outcomes in men with obstructive sleep apnoea-hypopnoea with or without treatment with continuous positive airway pressure: an observational study. Lancet. 2005 Mar 19-25;365(9464):1046-53. doi: 10.1016/S0140-6736(05)71141-7. PMID 15781100
- [Background] Campos-Rodriguez F, Pena-Grinan N, Reyes-Nunez N, De la Cruz-Moron I, Perez-Ronchel J, De la Vega-Gallardo F, Fernandez-Palacin A. Mortality in obstructive sleep apnea-hypopnea patients treated with positive airway pressure. Chest. 2005 Aug;128(2):624-33. doi: 10.1378/chest.128.2.624. PMID 16100147
- [Background] Grebe M, Eisele HJ, Weissmann N, Schaefer C, Tillmanns H, Seeger W, Schulz R. Antioxidant vitamin C improves endothelial function in obstructive sleep apnea. Am J Respir Crit Care Med. 2006 Apr 15;173(8):897-901. doi: 10.1164/rccm.200508-1223OC. Epub 2006 Jan 26. PMID 16439717
- [Background] Ip MS, Tse HF, Lam B, Tsang KW, Lam WK. Endothelial function in obstructive sleep apnea and response to treatment. Am J Respir Crit Care Med. 2004 Feb 1;169(3):348-53. doi: 10.1164/rccm.200306-767OC. Epub 2003 Oct 9. PMID 14551167
- [Background] Kato M, Roberts-Thomson P, Phillips BG, Haynes WG, Winnicki M, Accurso V, Somers VK. Impairment of endothelium-dependent vasodilation of resistance vessels in patients with obstructive sleep apnea. Circulation. 2000 Nov 21;102(21):2607-10. doi: 10.1161/01.cir.102.21.2607. PMID 11085964
- [Background] El Solh AA, Akinnusi ME, Baddoura FH, Mankowski CR. Endothelial cell apoptosis in obstructive sleep apnea: a link to endothelial dysfunction. Am J Respir Crit Care Med. 2007 Jun 1;175(11):1186-91. doi: 10.1164/rccm.200611-1598OC. Epub 2007 Feb 1. PMID 17272785
- [Background] Imadojemu VA, Gleeson K, Gray KS, Sinoway LI, Leuenberger UA. Obstructive apnea during sleep is associated with peripheral vasoconstriction. Am J Respir Crit Care Med. 2002 Jan 1;165(1):61-6. doi: 10.1164/ajrccm.165.1.2009062. PMID 11779731